CLINICAL TRIAL: NCT05626985
Title: Refinement and Validation of a Comprehensive Clinical Diagnostic Model (GAMAD) for Early Detection of Hepatocellular Carcinoma: A Multicenter, Prospective Study Protocol
Brief Title: Refinement and Validation of a Diagnostic Model (GAMAD) for Early Detection of Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: GAMAD
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: early detection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Hepatocellular Carcinoma patients: Blood samples are collected before liver resection.
  Interventions: Diagnostic Test: GAMAD
- Liver cirrhosis: The diagnosis of liver cirrhosis are based on triple-phase contrast enhanced computed tomography, magnetic resonance imaging.
  Interventions: Diagnostic Test: GAMAD
- Hepatitis: Patients with various hapatitis.
  Interventions: Diagnostic Test: GAMAD
- Benign tumor-like lesions: Benign hepatic tumors were diagnosed based on imaging findings and histological examinations after hepatic resection.
  Interventions: Diagnostic Test: GAMAD
- Healthy control: The healthy control group consist of people undergoing routine medical examination. Blood samples are collected.
  Interventions: Diagnostic Test: GAMAD

INTERVENTIONS:
Diagnostic Test: GAMAD — Blood samples are tested for tumor markers including PIVKA-II (DCP),AFP, ctDNA methylation and biochemical tests.

SUMMARY:
Most hepatocellular carcinoma (HCC) cases were at advanced stage when diagnosis established. This study is intended to establish a clinical diagnostic model GAMAD for early-stage HCC and evaluate the diagnostic efficiency the same time. This study is a multicenter prospective study. Participants including healthy control,HCC, liver cirrhosis, hepatitis and benign tumor-like lesions are consecutively recruited into the cohort. All the blood samples are collected before any treatments and will be tested in single center in order to decrease bias.

DETAILED DESCRIPTION:
GALAD score including age, sex, PIVKA-II(DCP), Alpha-fetoprotein (AFP) and alpha-fetoprotein L3 (AFP-L3), is a serum biomarker-based panel that can aid in early detection among patients with a high risk for liver cancer. While increasing studies showed the diagnostic accuracy of AFP-L3 was not as good as that of AFP or PIVKA-II, and AFP-L3 was not significant in the multivariable model. Thus, a model with better diagnostic accuracy and more suitable for Chinese patients is needed. Here, based on a multi-locus blood-based assay targeting circulating tumor DNA methylation, we aim to develop a novel diagnostic model--GAMAD (gender, age, methylation, AFP and DCP) and validate its performance among HCC patients and those at high risk of developing HCC,such as liver cirrhosis, hepatitis patients. This is a multicenter, observational, prospective study. After giving fully informed consent, the participants will undergo the regular treatment according to NCCN guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Establishing Diagnosis according to the European Association for the Study of Liver(EASL) criteria
* High risk group of developing HCC including liver cirrhosis and hepatitis under the confirmed diagnosis
* Able to provide sufficient and qualified blood samples for study tests
* No prior or undergoing cancer treatment (local or systematic)
* Able to provide a written informed consent

Exclusion Criteria:

* Obstructive jaundice patients
* Medical history of taking warfarin
* With other known malignant tumors or multiple primary tumors
* Patients with autoimmune diseases, genetic diseases, mental diseases/ disabilities and other diseases considered unsuitable for the study by the investigator
* During pregnancy or lactation
* Recipient of blood transfusion within 3 months prior to study blood draw
* Insufficient qualified blood sample for study test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients must have baseline evaluations performed prior to the study and must meet all inclusion and exclusion criteria. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent. The written informed consent must be obtained from the patient prior to enrollment. The following criteria apply to all patients enrolled onto the study unless otherwise specified
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
GAMAD | Day one
  Using GAMAD calculator model to obtain the score of each group.

SECONDARY OUTCOMES:
GALAD | Day one
  Using GALAD calculator to obtain the score of each group.
circulating tumor DNA methylation | Day one
  Using circulating tumor DNA methylation to obtain diagnostic value in pre-specified subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Tian Yang, Ph.D, Principal Investigator — Eastern Hepatobiliary Surgery Hospital; Guoyue Lv, Ph.D, Study Chair — The First Hospital of Jilin University; Fengmei Wang, Principal Investigator — Tianjin Third Central Hospital
Locations (3):
- China (3):
  - The First Hospital of Jilin University, Jilin
  - Eastern Hepatobiliary Surgery Hospital, Shanghai
  - Tianjin Third Central Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).

REFERENCES:
- [Background] Yang T, Xing H, Wang G, Wang N, Liu M, Yan C, Li H, Wei L, Li S, Fan Z, Shi M, Chen W, Cai S, Pawlik TM, Soh A, Beshiri A, Lau WY, Wu M, Zheng Y, Shen F. A Novel Online Calculator Based on Serum Biomarkers to Detect Hepatocellular Carcinoma among Patients with Hepatitis B. Clin Chem. 2019 Dec;65(12):1543-1553. doi: 10.1373/clinchem.2019.308965. Epub 2019 Oct 31. PMID 31672853
- [Background] Liu S, Sun L, Yao L, Zhu H, Diao Y, Wang M, Xing H, Lau WY, Guan M, Pawlik TM, Shen F, Xu M, Tong X, Yang T. Diagnostic Performance of AFP, AFP-L3, or PIVKA-II for Hepatitis C Virus-Associated Hepatocellular Carcinoma: A Multicenter Analysis. J Clin Med. 2022 Aug 29;11(17):5075. doi: 10.3390/jcm11175075. PMID 36079006
- [Derived] Yang T, Wang N, Wang F, Liu H, Shen F, Lv G. Refinement and validation of a comprehensive clinical diagnostic model (GAMAD) based on gender, age, multitarget circulating tumour DNA methylation signature and commonly used serological biomarkers for early detection of hepatocellular carcinoma: a multicentre, prospective observational study protocol. BMJ Open. 2023 Sep 18;13(9):e076467. doi: 10.1136/bmjopen-2023-076467. PMID 37723113